CLINICAL TRIAL: NCT02316613
Title: OLYMPE - Prospective Cohort Study on the Management of Patients With Relapsed Follicular Lymphoma
Brief Title: Prospective Observational Study on the Management of Patients With Relapsed or Refractory Follicular Lymphoma (OLYMPE)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML20248
Record Dates: First submitted 2014-11-28; First posted 2014-12-15 (Estimated); Results first posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-01

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- All Participants: Participants with histologically confirmed, refractory/relapsed cluster of differentiation-20 (CD20) positive follicular non-Hodgkin's lymphoma (grade IIII), whatever the first-line treatment was (chemotherapy and/or immunotherapy and/or radio-immunoconjugate and/or radiochemotherapy), and eligible for salvage treatment were observed for approximately 6 years. All participants received at least one cycle of rituximab (MabThera) during maintenance therapy or observation period.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab
  Other Names: MabThera®

SUMMARY:
This French national, multicenter, prospective, longitudinal, observational study will describe the treatment modalities of a cohort of patients with relapsed or refractory follicular non-Hodgkin's lymphoma, with evaluation of the cohort overall and according to the presence or not of MabThera® (rituximab) maintenance therapy. Actively participating physicians will enroll patients and collect therapeutic management data in a real-life setting up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age >/= 18 years)
* Presenting with WHO grade 1-3, CD20-positive follicular non-Hodgkin's lymphoma, histologically confirmed at initial diagnosis
* In relapse (or refractory) after at least one line of treatment, regardless of the nature of previous treatments (chemotherapy and/or immunotherapy and/or radioimmunoconjugate therapy and/or radiation+chemotherapy) and for whom a decision was made to give salvage therapy
* Having received oral and written information about the study and having raised no objections to electronic capture and processing of his/her personal data

Exclusion Criteria:

* Patient participating in a clinical trial evaluating a new, non-commercialized cancer treatment at the time of inclusion
* Follicular lymphoma presenting with a transformation to diffuse large cell non-Hodgkin's lymphoma
* First line treatment with radiotherapy alone
* Initial abstention from treatment (decision to not treat the progression at the time of inclusion in the OLYMPE study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment of approximately 90 physicians who treat patients with follicular non-Hodgkin's lymphoma to actively participate in this observational study. Patients with relapsed or refractory follicular non-Hodgkin's lymphoma (World Health Organization grade 1-3) and requiring treatment are to be enrolled prospectively. Subgroup of interest: patients receiving MabThera® (rituximab) maintenance therapy.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2007-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Neuilly-sur-Seine, France

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 260 participants, 5 were excluded as no data available and duplicate cases (N=255; safety population) and 14 were excluded as other selection criteria not met (N=241; overall population).
Groups:
- All Participants: Participants with histologically confirmed, refractory/relapsed cluster of differentiation-20 (CD20) positive follicular non-Hodgkin's lymphoma (grade IIII), whatever the first-line treatment was (chemotherapy and/or immunotherapy and/or radio-immunoconjugate and/or radiochemotherapy), and eligible for salvage treatment were observed for approximately 6 years.
Period: Overall Study
Arm/Group | All Participants
Started | 260
Safety Population | 255
Overall Population | 241
Completed | 156
Not Completed | 104
Not completed — Death | 63
Not completed — Lost to Follow-up | 9
Not completed — Lymphoma transformation | 2
Not completed — Participant moved/changed medical team | 11
Not completed — No data and duplicate cases | 5
Not completed — Did not met selection criteria | 14

BASELINE CHARACTERISTICS:
Population: Overall population: All the participants (except duplicate cases and participants without data available) meeting all the inclusion/exclusion criteria were included.
Groups:
- All Participants: Participants with histologically confirmed, refractory/relapsed CD2 0-positive follicular non-Hodgkin's lymphoma (grade IIII), whatever the first-line treatment was (chemotherapy and/or immunotherapy and/or radio-immunoconjugate and/or radiochemotherapy), and eligible for salvage treatment were observed for approximately 6 years.
Arm/Group | All Participants
Number analyzed (Participants) | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 131

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Modalities of the Therapeutic Decision Before First Study Induction Treatment Phase
Description: At study inclusion, the therapeutic management of participants was decided by either "pluri-disciplinary consultation meeting," "Only the physician in charge of the participant," "Discussion between physicians," or "Punctual consultation of an external physician." Percentage of participants with each of these modalities of therapeutic decision was reported.
Time Frame: Baseline
Population: Overall population: All the participants (except duplicate cases and participants without data available) meeting all the inclusion/exclusion criteria were included. Number of participants analyzed = participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 238
percentage of participants
  Pluri-disciplinary consultation meeting | 81.9
  Only the physician in charge of the participants | 8.4
  Discussion between physicians | 6.3
  Punctual consultation of an external physician | 3.4

2. Secondary Outcome: Percentage of Participants With Last Induction Treatment Response
Description: Last Induction treatment response: the last response assessment over the first study induction treatment (complete response [CR]: complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy; CR unconfirmed: CR along with regression in lymph node mass by more than [>]75% in the sum of the products of greatest diameters [SPD]; Partial Response [PR]: greater than or equal to [>=] 50% decrease in SPD of 6 largest dominant nodes or nodal masses; Progression was 1 of the following: 1) lymphadenopathy; 2) a >=50% increase in previously noted or new appearance of hepato/splenomegaly; 3) >=50% increase in blood lymphocyte count with at least 5000 B lymphocytes/μL; 4) transformation to Richter's syndrome; or 5) occurrence of cytopenia; Stable disease [SD]: absence of necessary criteria to achieve CR or PR, but no advancement to progression) was described at the end of first study induction.
Time Frame: Induction Phase: 18.7 months
Population: Overall population: All the participants (except duplicate cases and participants without data available) meeting all the inclusion/exclusion criteria were included. Number of participants analyzed (N)=number of participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Groups:
- All Participants: Participants with histologically confirmed, refractory/relapsed CD20-positive follicular non-Hodgkin's lymphoma (grade IIII), whatever the first-line treatment was (chemotherapy and/or immunotherapy and/or radio-immunoconjugate and/or radiochemotherapy), and eligible for salvage treatment.
Arm/Group | All Participants
Number analyzed (Participants) | 227
percentage of participants
  Complete response | 38.3
  Complete response not confirmed | 11.5
  Partial response >=50% | 31.7
  Partial response <50% | 6.2
  Stability | 5.3
  Progression | 7.0

3. Secondary Outcome: Percentage of Participants With Number of Disease Progressions
Description: Participants with at least one disease progression after the first study induction period were reported.
Time Frame: Up to 6 years
Population: Overall population: All the participants (except duplicate cases and participants without data available) meeting all the inclusion/exclusion criteria were included. Number of participants analyzed= those participants who entered in maintenance/observation after the first induction and before the first disease progression over the study.
Measure: Number; unit: percentage of participants
Groups:
- Without MabThera: Treatment without MabThera was defined as the absence of MabThera administration during maintenance therapy or observation period.
- MabThera as Maintenance Therapy: Treatment with MabThera was defined as the administration of at least one cycle of MabThera during maintenance therapy or observation period.
Arm/Group | Without MabThera | MabThera as Maintenance Therapy
Number analyzed (Participants) | 74 | 127
percentage of participants
  Number of disease progressions: 0 | 52.7 | 68.5
  Number of disease progressions: 1 | 39.22 | 22.0
  Number of disease progressions: 2 | 6.8 | 6.3
  Number of disease progressions: 3 | 1.4 | 2.4
  Number of disease progressions: 4 | 0.0 | 0.8

4. Secondary Outcome: Percentage of Participants With Disease Characteristics at First Study Disease Progression
Description: Disease characteristics included (tumor burden, measured from whole body computed tomography (CT) scan. Groupe d'Etudes des Lymphomes Folliculaires (GELF) criteria defined as parameters to initiate treatment in participants with untreated follicular lymphoma, grade 1,2,or 3A; having just one of the criteria justified treatment: 1. involvement of >=3 nodal sites, each with diameter of >=3 centimeter(cm); 2. any nodal/extranodal tumor mass with diameter of >=7cm; 3. B symptoms (temperature >=38 degrees celsius or night sweats or weight loss >10% over past 6 months); 4. splenomegaly; 5. pleural effusion/peritoneal ascites; 6. cytopenia (leukocytes <1×10^9 and/or platelets <100×10^9/L. One participant could present with more than 1 GELF criterion. Ann Arbor staging was used as staging system for lymphomas (Stage I to IV); stage depended upon the place where malignant tissue was located (through biopsy, CT scan, or positron emission tomography) and on systemic symptoms due to lymphoma).
Time Frame: Up to 6 years
Population: Overall population: All the participants (except duplicate cases and participants without data available) meeting all the inclusion/exclusion criteria were included. Number of participants analyzed= participants with at least one disease progression over the study period. n=number of evaluable participant for each disease characteristics.
Measure: Number; unit: percentage of participants
Arm/Group | Without MabThera | MabThera as Maintenance Therapy
Number analyzed (Participants) | 35 | 39
percentage of participants
  Tumor burden: Data not available (n=32, 38) | 3.1 | 5.3
  Tumor burden: High (n=32, 38) | 50.0 | 42.1
  Tumor burden: Low (n=32, 38) | 46.9 | 52.6
  GELF criteria: at least 3 nodal sites (n=32, 38) | 12.5 | 21.1
  GELF criteria: Any nodal/extra-nodal mass(n=32,38) | 12.5 | 18.4
  GELF criteria: B symptoms (n=32, 38) | 12.5 | 0.0
  GELF criteria: Splenomegaly (n=32, 38) | 9.4 | 2.6
  GELF criteria: Pleural/ascites effusion (n=32, 38) | 6.3 | 7.9
  GELF criteria: Cytopenia (n=32, 38) | 6.3 | 0.0
  GELF criteria: None (n=32, 38) | 46.9 | 52.6
  GELF criteria: Not available (n=32, 38) | 3.1 | 5.3
  Ann-Arbor stage I (n=35, 39) | 11.4 | 15.4
  Ann-Arbor stage II (n=35, 39) | 14.3 | 10.3
  Ann-Arbor stage III (n=35, 39) | 14.3 | 15.4
  Ann-Arbor stage IV (n=35, 39) | 37.1 | 33.3
  Ann-Arbor stage data not available (n=35, 39) | 17.1 | 23.1
  Ann-Arbor stage not assessable (n=35, 39) | 5.7 | 2.6

5. Secondary Outcome: Progression Free Survival (PFS)
Description: The PFS was defined as the time from the date of first induction treatment over the study (first treatment administration of first cycle) to the date of first disease progression or participants death or date of lymphoma transformation diagnosis.
Time Frame: Up to 6 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Groups:
- All Participants: Participants with histologically confirmed, refractory/relapsed CD20-positive follicular non-Hodgkin's lymphoma (grade IIII), whatever the first-line treatment was (chemotherapy and/or immunotherapy and/or radio-immunoconjugate and/or radiochemotherapy), and eligible for salvage treatment were observed for approximately 6 years.
Arm/Group | All Participants
Number analyzed (Participants) | 241
months | 44.4 [33.9 to 54.7]

6. Secondary Outcome: Time to Next Treatment
Description: Time to next treatment was calculated from the date of the end of first induction treatment administration over the study to the date of the start of next treatment after disease progression.
Time Frame: Up to 6 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Participants
Number analyzed (Participants) | 241
months | NA [NA to NA] — Median time to next treatment and 95% confidence interval (CI) were not estimated due to insufficient (<50%) participants with the event of interest.

7. Secondary Outcome: Overall Survival (OS)
Description: The overall survival was defined as the time from the date of first induction treatment administration over the study to the date of participants' death or early study withdrawal. OS was calculated using Kaplan-Meier method.
Time Frame: Up to 6 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Participants
Number analyzed (Participants) | 241
months | NA [NA to NA] — Median time to next treatment and 95% CI were not estimated due to insufficient (<50%) participants with the event of interest.

8. Secondary Outcome: Number of Participants Who Used MabThera
Time Frame: Up to Induction phase (18.7 months), Maintenance phase/observation phase (67.8 months)
Population: All the participants (except duplicate cases and participants without data available) meeting all the inclusion/exclusion criteria were included.
Measure: Number; unit: participants
Groups:
- All Participants: Participants with histologically confirmed, refractory/relapsed CD20-positive follicular non-Hodgkin's lymphoma (grade IIII), whatever the first-line treatment was (chemotherapy and/or immunotherapy and/or radio-immunoconjugate and/or radiochemotherapy), and eligible for salvage treatment were observed for approximately 6 years. Participants who received MabThera treatment over the first study induction period was reported.
- MabThera as Maintenance Therapy: Treatment with MabThera was defined as the administration of at least one cycle of MabThera during maintenance therapy or observation period. Participants who received MabThera maintenance therapy after the first study induction was reported.
Arm/Group | All Participants | MabThera as Maintenance Therapy
Number analyzed (Participants) | 241 | 127
participants
  At least one cycle of MabThera | 230 | 127
  All cycles with MabThera (monotherapy/combination) | 205 | 127
  At least one cycle of MabThera as monotherapy | 89 | 125
  All cycles with MabThera as monotherapy | 51 | 124
  At least one cycle of MabThera in combination | 178 | 2
  All cycles with MabThera in combination | 119 | 1

9. Primary Outcome: Percentage of Participants With Treatments Prescribed Over the First Study Induction Phase
Description: Over the first treatment induction period, participants received following therapies for the treatment of refractory/relapsed follicular non-Hodgkin's lymphoma: chemotherapy combined with MabThera, chemotherapy alone, MabThera monotherapy, and stem cell transplantation, radio-immunotherapy, or radiation therapy combined with any other treatment. Study induction treatment phase consists total of three visits (one before the first cycle, one halfway through therapy and one after the last cycle to evaluate response). Induction treatment duration ranged between <3 months to >6 months. Each participants may received more than one therapy.
Time Frame: Induction Phase: 18.7 months
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 241
percentage of participants
  Chemotherapy plus MabThera | 47.7
  MabThera as monotherapy | 21.2
  Stem Cells Transplantation | 19.5
  Radio-immunotherapy | 11.2
  Chemotherapy alone | 2.9
  Radiation therapy | 2.5

10. Primary Outcome: Percentage of Participants With Chemotherapies Prescribed Over the First Study Induction Phase
Description: Over the first study induction phase, participants received the following chemotherapy: regimen including fludarabine; regimen including aracytine - platinum salts; cyclophosphamide/hydroxydaunorubicin/oncovin/prednisone (CHOP-like); cyclophosphamide/vincristine/prednisone (CVP); regimen including ifosfamide - etoposide; and other chemotherapy. One participant could receive more than one type of chemotherapy over the first treatment induction period.
Time Frame: Induction Phase: 18.7 months
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 122
percentage of participants
  Regimen including fludarabine | 45.9
  Regimen including aracytine - platinum salts | 44.3
  CHOP-like | 32.0
  CVP | 13.1
  Regimen including ifosfamide - etoposide | 10.7
  Other chemotherapy | 23.8

11. Primary Outcome: Percentage of Participants With MabThera as Maintenance Therapy
Description: During the maintenance period participants received four weekly infusion of MabThera.
Time Frame: Maintenance/observation Phase: 67.8 months
Population: Overall population: All the participants (except duplicate cases and participants without data available) meeting all the inclusion/exclusion criteria were included. Number of participants analyzed= those who entered in maintenance/observation after the first induction and before the first disease progression over the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 201
percentage of participants | 63.2 [56.5 to 69.9]

12. Primary Outcome: Percentage of Participants With MabThera Maintenance Therapy and at Least One Observation Phase
Description: After study induction period (three visits) participants entered into either of two periods: 1. period of maintenance with MabThera followed by observation or 2. period of observation/maintenance without MabThera, followed by maintenance with MabThera.
Time Frame: Maintenance/observation Phase: 67.8 months
Population: Overall population: All the participants (except duplicate cases and participants without data available) meeting all the inclusion/exclusion criteria were included. Number of participants analyzed = those who received at least one MabThera infusion over the maintenance therapy period.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 127
percentage of participants
  Maintenance with MabThera followed by observation | 70.9
  Observation followed by maintenance with MabThera | 1.6
  Only maintenance therapy | 27.6

13. Primary Outcome: Duration of MabThera Maintenance Therapy When Associated With Observation
Description: Duration of MabThera maintenance therapy was calculated from the end of induction period to the day before the first disease progression over the study (or to the date of last participant information if no disease progression until the end of the participant follow-up). Disease progression was based on the followings: Eastern Cooperative Oncology Group performance status; presence of B symptoms (fever 38°C in absence of infection for more than 8 days, night sweats, weight loss exceeding 10% in 6 months); evaluation of tumor mass (Groupe d'Etudes des Lymphomes Folliculaires criteria); number of nodal sites; number and location of extranodal sites; Ann-Arbor stage (I to IV); any histological documentation: type of biopsy (nodal, extranodal, bone marrow); histological type (progression of follicular non-Hodgkin's lymphomas or transformation); latest available hemoglobin, neutrophils, normal or leukemic lymphocytes, platelets, lactate dehydrogenase, and total gamma globulins level.
Time Frame: Maintenance/observation Phase: 67.8 months
Population: Overall population: All the participants (except duplicate cases and participants without data available) meeting all the inclusion/exclusion criteria were included. Number of participants analyzed = those who received at least one infusion of MabThera and completed maintenance therapy with MabThera when associated with observation period.
Measure: Median (Full Range); unit: months
Arm/Group | All Participants
Number analyzed (Participants) | 92
months | 24.5 [3.2 to 37.7]

14. Primary Outcome: Percentage of Participants With Prescription of Injection Prophylaxis
Description: Participants was prescribed with either of the following infection prophylaxis treatment: anti-pneumocystosis agents, antiviral agents, or immunoglobulins.
Time Frame: Maintenance/observation Phase: 67.8 months
Population: Overall population: All the participants (except duplicate cases and participants without data available) meeting all the inclusion/exclusion criteria were included. Number of participants analyzed=all participants having had maintenance/observation period before the first study disease progression.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 201
percentage of participants | 39.3

15. Primary Outcome: Percentage of Participants With Injection Prophylaxis Treatment
Description: Participants received anti-pneumocystosis agents, antiviral agents, or immunoglobulins as infection prophylaxis. One participant could receive more than one infection prophylaxis treatment.
Time Frame: Maintenance/observation Phase: 67.8 months
Population: Overall population: All the participants (except duplicate cases and participants without data available) meeting all the inclusion/exclusion criteria were included. Number participants analyzed= all participants having had maintenance/observation period before the first study disease progression and received infection prophylaxis treatment.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 79
percentage of participants
  Anti-pneumocystosis agent | 65.8
  Antiviral agents | 83.5
  Immunoglobulins | 26.9

16. Primary Outcome: Percentage of Participants With Modalities of the Therapeutic Decision at First Study Disease Progression
Description: The therapeutic management of participants was decided by either "pluri-disciplinary consultation meeting," "Only the physician in charge of the participant," "Discussion between physicians," or "Punctual consultation of an external physician." Percentage of participants with each of these modalities of therapeutic decision was reported.
Time Frame: Up to 6 years
Population: Overall population: All the participants (except duplicate cases and participants without data available) meeting all the inclusion/exclusion criteria were included. Number of participants analyzed= participants with at least one disease progression over the study period.
Measure: Number; unit: percentage of participants
Arm/Group | Without MabThera | MabThera as Maintenance Therapy
Number analyzed (Participants) | 35 | 40
percentage of participants
  Pluri-disciplinary consultation meeting | 80.0 | 67.5
  Only physician in charge of the participant | 17.1 | 20.0
  Discussion between physicians | 2.9 | 10.0
  Punctual consultation with an external physician | 0.0 | 2.5

17. Primary Outcome: Number of Participants With Therapeutic Management After the First Study Disease Progression
Description: After the first disease progression the participants received chemotherapy, immunotherapy, radio immunotherapy, stem cell transplantation, or radiation therapy for therapeutic management of the refractory/relapsed follicular non-Hodgkin's lymphoma. One participant could receive more than one type of treatment after the first study disease progression.
Time Frame: Up to 6 years
Population: as for outcome 16
Measure: Number; unit: participants
Arm/Group | Without MabThera | MabThera as Maintenance Therapy
Number analyzed (Participants) | 35 | 40
participants
  Missing | 2 | 4
  Chemotherapy | 24 | 29
  Immunotherapy | 24 | 27
  Radio immunotherapy | 0 | 4
  Stem cell transplantation | 7 | 7
  Radiation therapy | 6 | 5

18. Secondary Outcome: MabThera Regimen: Dose of MabThera
Description: All participants who received MabThera treatment before the first disease progression were reported.
Time Frame: Up to Induction phase (18.7 months), Maintenance phase/observation phase (67.8 months)
Population: All the participants (except duplicate cases and participants without data available) meeting all the inclusion/exclusion criteria were included. Number of participants analyzed= participants who received at least one cycle of MabThera and available with valid data for this outcome.
Measure: Mean (Standard Deviation); unit: milligram (mg)
Groups:
- All Participants: Participants with histologically confirmed, refractory/relapsed CD20-positive follicular non-Hodgkin's lymphoma (grade IIII), whatever the first-line treatment was (chemotherapy and/or immunotherapy and/or radio-immunoconjugate and/or radiochemotherapy), and eligible for salvage treatment were observed for approximately 6 years. Participants who received treatment with MabThera over the first study induction period was reported.
- MabThera as Maintenance Therapy: Treatment with MabThera was defined as the administration of at least one cycle of MabThera during maintenance therapy or observation period. Participants who received treatment with MabThera after the first study induction period was reported.
Arm/Group | All Participants | MabThera as Maintenance Therapy
Number analyzed (Participants) | 216 | 125
milligram (mg) | 661.25 (92.94) | 671.15 (111.05)

19. Secondary Outcome: MabThera Regimen: Infusion Duration
Time Frame: Up to Induction phase (18.7 months), Maintenance phase/observation phase (67.8 months)
Population: All the participants (except duplicate cases and participants without data available) meeting all the inclusion/exclusion criteria were included. Number of participants analyzed= participants who received at least one cycle of MabThera and available with valid data.
Measure: Mean (Standard Deviation); unit: minutes (mn)
Arm/Group | All Participants | MabThera as Maintenance Therapy
Number analyzed (Participants) | 199 | 103
minutes (mn) | 168.60 (64.74) | 150.25 (60.09)

20. Secondary Outcome: MabThera Regimen: Number of Cycles of MabThera
Time Frame: Up to Induction phase (18.7 months), Maintenance phase/observation phase (67.8 months)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: number of cycles
Arm/Group | All Participants | MabThera as Maintenance Therapy
Number analyzed (Participants) | 230 | 125
number of cycles | 4.8 (1.9) | 7.6 (3.2)

21. Secondary Outcome: MabThera Regimen: Time Between Cycles
Time Frame: Up to Induction phase (18.7 months), Maintenance phase/observation phase (67.8 months)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: days
Arm/Group | All Participants | MabThera as Maintenance Therapy
Number analyzed (Participants) | 222 | 119
days | 23.79 (12.04) | 80.60 (20.69)

22. Secondary Outcome: Percentage of Participants With Discontinuations and Modifications of MabThera During Maintenance Phase
Time Frame: Maintenance phase : 67.8 months
Population: All the participants (except duplicate cases and participants without data available) meeting all the inclusion/exclusion criteria were included. Number of participants analyzed= participants who received at least one MabThera infusion over the maintenance therapy period. n=number of evaluable participants for each category.
Measure: Number; unit: percentage of participants
Arm/Group | MabThera as Maintenance Therapy
Number analyzed (Participants) | 123
percentage of participants
  Treatment discontinuation: Yes (n=123) | 6.5
  Treatment discontinuation: No (n=123) | 93.5
  At least 1 dose modification: Yes (n=121) | 41.3
  At least 1 dose modification: No (n=121) | 58.7
  At least 1 duration modification: Yes (n=121) | 36.4
  At least 1 duration modification: No (n=121) | 63.6
  Number (No.) of dose modifications: 0 (n=121) | 58.7
  No. of dose modifications: 1 (n=121) | 17.4
  No. of dose modifications: 2 (n=121) | 10.7
  No. of dose modifications: 3 (n=121) | 5.8
  No. of dose modifications: 4 (n=121) | 4.1
  No. of dose modifications: 5 (n=121) | 2.5
  No. of dose modifications: 6 (n=121) | 0.8
  No. of infusion duration modifications: 0 (n=121) | 63.6
  No. of infusion duration modifications: 1 (n=121) | 10.7
  No. of infusion duration modifications: 2 (n=121) | 5.8
  No. of infusion duration modifications: 3 (n=121) | 4.1
  No of infusion duration modifications: 4 (n=121) | 3.3
  No. of infusion duration modifications: 5 (n=121) | 5.0
  No. of infusion duration modifications: 6 (n=121) | 1.7
  No. of infusion duration modifications: 7 (n=121) | 2.5
  No. of infusion duration modifications: 8 (n=121) | 2.5
  No. of infusion duration modifications: 9 (n=121) | 0.8

23. Secondary Outcome: Function Assessment of Chronic Illness Therapy-General (FACT-G) With Lymphoma-Specific Additional Concerns Subscale (Lym) Total Score
Description: The FACT-G with Lymphoma-Specific Additional Concerns Subscale (Lym) total score was calculated by adding the score obtained on the FACT-G (physical well-being, scored 0-28; social well-being, scored 0-28; functional well-being, scored 0-28; emotional well-being, scored 0-24), to the score obtained on the LYM subscale (15 items; responses to each item range from 0, "Not at all" to 4, "Very much"). Total score ranges from 0 to 168. Higher scores indicated a better participant-reported outcome/quality of life over the past week when responding to the items.
Time Frame: Up to 6 years (assessed at start, mid and end of induction [induction: 18.7 months], at each infusion during maintenance [maintenance phase: 67.8 months], and at disease progression [maximum up to 6 years])
Population: All the participants (except duplicate cases and participants without data available) meeting all the inclusion/exclusion criteria were included. n=number of evaluable questionnaires for each category.
Measure: Mean (Standard Deviation); unit: score on scale
Units Other Than Participants: Total number of assessable questionnaire
Arm/Group | All Participants
Number analyzed (Participants) | 241
Number analyzed (Total number of assessable questionnaire) | 666
score on scale
  Physical well-being (n=661) | 22.14 (4.99)
  Social well-being (n=660) | 17.67 (5.31)
  Emotional well-being (n=664) | 17.30 (4.46)
  Functional well-being (n=659) | 15.32 (5.69)
  Other worrying participants (n=662) | 45.92 (8.88)
  Global score (n=663) | 118.11 (23.09)

24. Secondary Outcome: Number and Type of Hospitalization Associated With MabThera Perfusion
Description: Number and type of hospitalization (a day hospitalization, short-lasting hospitalization, and short-stay hospitalization) was reported.
Time Frame: Up to 6 years
Population: as for outcome 8
Measure: Number; unit: hospitalizations
Units Other Than Participants: cycles with MabThera
Groups:
- First Induction: During the induction period participants received either MabThera monotherapy, MabThera combination therapy (chemotherapy and at least one cycle with MabThera), or all cycles performed without MabThera administration.
- Maintenance Therapy: During maintenance therapy the participants received or did not received treatment with the MabThera.
Arm/Group | First Induction | Maintenance Therapy
Number analyzed (Participants) | 241 | 201
Number analyzed (cycles with MabThera) | 1035 | 951
hospitalizations
  A day hospitalization | 727 | 934
  Short-lasting hospitalization | 308 | 15
  Short-stay hospitalization | 0 | 2

ADVERSE EVENTS:
Time Frame: Up to 6 years
Description: Safety population (all participants, except duplicate cases and participants without data available) included 255 participants, here data for 243 participants is reported as 12 participants data were not available (participants without available follow-up for adverse effects).
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 94/243
Other Adverse Events (participants affected / at risk) | 134/243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=243)
Lung infection (Infections and infestations) | 15
Urinary tract infection (Infections and infestations) | 5
Bacteraemia (Infections and infestations) | 4
Bronchopulmonary aspergillosis (Infections and infestations) | 3
Pneumocystis jiroveci pneumonia (Infections and infestations) | 3
Septic shock (Infections and infestations) | 3
Herpes zoster (Infections and infestations) | 2
Abdominal infection (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Aspergillosis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Conjunctivitis infective (Infections and infestations) | 1
Haemophilus infection (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 1
Onychomycosis (Infections and infestations) | 1
Oropharyngeal candidiasis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1
Pyelonephritis acuts (Infections and infestations) | 1
Reiter's syndrome (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Ureapasma infection (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer metastic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hair follicle tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Refractory cytopenia with multilineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pyrexia (General disorders) | 7
Disease progression (General disorders) | 6
Death (General disorders) | 3
General physical health deterioration (General disorders) | 3
Chest pain (General disorders) | 1
Fatigue (General disorders) | 1
Hypothermia (General disorders) | 1
Multi-organ failure (General disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Agranulocytosis (Blood and lymphatic system disorders) | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1
Myocardial infarction (Cardiac disorders) | 3
Cardiac disorder (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Abdominal adhesions (Gastrointestinal disorders) | 1
Colitits ulcerative (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Aneurysm (Vascular disorders) | 1
Arterial stenosis (Vascular disorders) | 1
Cerebrovascular accident (Vascular disorders) | 1
Ischaemic stroke (Vascular disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
Hypogammaglobulinaemia (Immune system disorders) | 3
Fall (Injury, poisoning and procedural complications) | 1
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Encephalopathy (Nervous system disorders) | 2
Balance disorder (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Blindness (Eye disorders) | 1
Optic neuropathy (Eye disorders) | 1
CD4 lymphocytes decreased (Investigations) | 1
Inguinal hernia repair (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=243)
Bronchitis (Infections and infestations) | 47
Herpes zoster (Infections and infestations) | 14
Pharyngitis (Infections and infestations) | 12
Sinusitis (Infections and infestations) | 12
Pyrexia (General disorders) | 49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.